CLINICAL TRIAL: NCT05552196
Title: A Phase 1, Open-label, Parallel-group Study to Assess the Effect of Steady-state Carbamazepine on the Pharmacokinetics of Ponesimod in Healthy Adult Participants
Brief Title: A Study of Ponesimod in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109254; 2022-000502-97 (EudraCT Number); 67896153MSC1001 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — ponesimod; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: Ponesimod (Experimental): Participants will receive up-titrated Ponesimod orally once daily from Day 1 to Day 15.
  Interventions: Drug: Ponesimod
- Treatment B: Ponesimod + Carbamazepine (Experimental): Participants will receive up-titrated Carbamazepine from Day 1 to Day 7 and from Day 23 to Day 26. Participants will also receive up-titrated Ponesimod and Carbamazepine from Day 8 to Day 22.
  Interventions: Drug: Ponesimod; Drug: Carbamazepine

INTERVENTIONS:
Drug: Ponesimod — Ponesimod tablet will be administered orally.
  Other Names: JNJ-67896153; ACT-128800; Ponvory
Drug: Carbamazepine — Carbamazepine tablet will be administered orally.
  Other Names: Tegretol
  Arms: Treatment B: Ponesimod + Carbamazepine

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state carbamazepine (CBZ; a strong pregnane X receptor [PXR] agonist) on the pharmacokinetics (PK) of ponesimod following a gradual up-titration regimen in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between (BMI) 18-30 kilograms per meter square (kg/m^2)
* Willing and able to adhere to the prohibitions and restrictions.
* Female participants with negative pregnancy test.
* Women of childbearing potential (WOCBP) must use 2 methods of contraception.
* Healthy on the basis of physical examination (including neurological examination and skin examination), Columbia suicide severity rating scale questionnaire (C-SSRS) questionnaire, ophthalmological examination, medical history, vital signs, and 12-lead electrocardiogram (ECG).
* Positive varicella zoster virus (VZV).

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 60 milliliter per minute [mL/min]), thyroid disease, neurologic or psychiatric disease, confirmed or suspected macular edema, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results.
* Contraindications to the use of Carbamazepine (CBZ) as per local prescribing information
* Any immunosuppressive treatment within 6 weeks before first study drug administration.
* Lymphopenia (less than 1,000 cells per microliter).
* Received an investigational drug or used an invasive investigational medical device within 30 days before the first study drug intake or received a biological product within 3 months or 5 half-lives (whichever is longer) before the first study drug intake, or is currently enrolled in an investigational study.
* Lack of good/reasonable venous access.
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Treatment A: Cmax is the maximum Observed Plasma Concentration (Cmax) of Ponesimod | Pre dose up to 120 hours post dose on Day 15
  Cmax is the maximum observed plasma concentration of Ponesimod.
Treatment A: Area Under The Plasma Concentration-time Curve of Ponesimod From Time 0 to 24 Hours Post Dose (AUC [0-24h]) | Pre dose up to 120 hours post dose on Day 15
  AUC (0-24h) is the plasma concentration-time curve of Ponesimod from time 0 to 24 hours post dose, calculated by linear-linear trapezoidal summation.
Treatment B: Cmax is the maximum Observed Plasma Concentration (Cmax) of Ponesimod | Pre dose up to 120 hours post dose on Day 22
  Cmax is the maximum observed plasma concentration of Ponesimod.
Treatment B: Area Under The Plasma Concentration-time Curve of Ponesimod From Time 0 to 24 Hours Post Dose (AUC [0-24h]) | Pre dose up to 120 hours post dose on Day 22
  AUC (0-24h) is the plasma concentration-time curve of Ponesimod from time 0 to 24 hours post dose, calculated by linear-linear trapezoidal summation.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to Day 27
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Total Lymphocyte Count | Treatment A: Day 1 (Baseline) and Day 16; Treatment B: Day 1 (Baseline) and Day 23
  Total lymphocyte count will be reported.
Percentage Change in Lymphocytes From Baseline | Treatment A: Baseline and Day 16, Treatment B: Baseline and Day 23
  Percentage change in lymphocytes from baseline will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency